CLINICAL TRIAL: NCT03262610
Title: Expanded-access for the Use of Setmelanotide in a Single Patient With Partial Lipodystrophy (LD) Associated With Leptin Deficiency and Multiple Autoimmune Diseases
Brief Title: Setmelanotide in a Single Patient With Partial Lipodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-493-019
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Hypertriglyceridemia; Obesity
MeSH Terms: conditions — Hypertriglyceridemia; Obesity | interventions — setmelanotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Setmelanotide daily subcutaneous injection (Experimental): Up to 18 weeks setmelanotide treatment.
  Interventions: Drug: Setmelanotide

INTERVENTIONS:
Drug: Setmelanotide — daily subcutaneous injection
  Other Names: RM-493

SUMMARY:
The objective of this single patient study is to assess the safety and efficacy of setmelanotide as a treatment of severe metabolic abnormalities resulting from LD, especially refractory hypertriglyceridemia leading to recurrent bouts of pancreatitis.

DETAILED DESCRIPTION:
This is a single-patient study to assess the safety and efficacy of setmelanotide in a unique patient with partial LD and severe metabolic abnormalities, most notably refractory hypertriglyceridemia leading to recurrent pancreatitis despite ongoing plasmapheresis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Ability to comply with visits and procedures required by program.
3. Has physician-confirmed partial lipodystrophy and the following characteristics:

   * Has atypical lipodystrophy.
   * Has presence of neutralizing antibody to metreleptin
   * Patient has life threatening hypertriglyceridemia and has had >8 episodes of pancreatitis, requiring weekly plasmapheresis
   * Has Type 1 diabetes mellitus with HbA1c > 10%.
4. Female, under the age of 18 years

Exclusion Criteria:

1. Diagnosis of schizophrenia, bipolar disorder, personality disorder or other Diagnostic and Statistical Manual of Mental Disorders (DSM-III) disorders that the investigator believes will interfere significantly with study compliance. Neurocognitive disorders affecting ability to consent will not be disqualifying as long as an appropriate guardian able to give consent has been appointed.
2. History or close family history (parents or siblings) of skin cancer or melanoma, or patient history of ocular-cutaneous albinism.
3. Significant dermatologic findings relating to melanoma or pre-melanoma skin lesions, determined as part of a screening comprehensive skin evaluation performed by a qualified dermatologist.
4. Significant hypersensitivity to study drug.
5. Inability to comply with QD injection regimen.

Ages: 15 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — This is a single patient study
Enrollment: 1 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Fasting Triglycerides (TG) levels | 12 to 20 weeks
  The mean change from baseline in fasting triglycerides after setmelanotide treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Shapiro, M.D., Ph.D., Study Chair — Chief Medical Officer, Rhythm Pharmaceuticals, Inc
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States